CLINICAL TRIAL: NCT02362919
Title: Determinants of Vaccine Response to Influenza Vaccination Among Individuals Over 65 Years of Age - a Population-based Study
Brief Title: Influenza Vaccination Among the Elderly Individuals
Status: Completed | Type: Observational
Sponsor: Helmholtz Centre for Infection Research (Other)
Collaborators: Clinical Research Center, Hannover, Germany (Unknown); Hannover Unified Biobank, Hannover, Germany (Unknown); Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 1100359
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Influenza vaccination; Elderly individuals; Prospective cohort study; response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A cohort of elderly individuals: A cohort of elderly individuals between 65 and 80 years of age were vaccinated with Fluad, a seasonal inactivated trivalent adjuvanted influenza vaccine. Blood samples before (day 0) and at days 1/3, 7,21 and 70 after vaccination were collected.

SUMMARY:
The aims of the study are to a) identify individuals with a poor response to influenza vaccination and b) identify factors associated with a poor response to influenza vaccination.

DETAILED DESCRIPTION:
This is a population-based prospective cohort study. Potential participants, males and females between 65 and 80 years of age, were selected randomly through the resident registration office in Hannover city, Germany and invited with a personalized letter to participate in the study.

Initially, a blood sample (40 ml) will be drawn from each participant (day 0). Furthermore, participants will be vaccinated against influenza with FLUAD 2014/2015. FLUAD is a trivalent, surface antigen, inactivated influenza virus vaccine adjuvanted with MF59C.1. Additional five blood samples will be collected during the study period of four months (at days 3, 7, 21, 70 and 130). Information about current and past infections, chronic diseases and basic sociodemographic data will be collected through a self-administered questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 65 and 80 years of age

Exclusion Criteria:

* Individuals with a known hypersensitivity to any of the excipients and to eggs, chicken Protein, kanamycin and neomycin sulphate, formaldehyde, and cetyltrimethylammonium bromide
* Individuals, who have an acute infection during the visit at the study Center
* Individuals with cognitive impairment
* Individuals already vaccinated with influenza vaccination in the influenza season 2014/15

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Males and females aged 65 and 80 years from the general population
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Serological evidence of vaccine response to influenza vaccination | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pessler, PD Dr., Principal Investigator — Twincore Centre for Experimental and Clinical Infection Research, Hannover, Germany

REFERENCES:
- [Derived] Akmatov MK, Riese P, Trittel S, May M, Prokein J, Illig T, Schindler C, Guzman CA, Pessler F. Self-reported diabetes and herpes zoster are associated with a weak humoral response to the seasonal influenza A H1N1 vaccine antigen among the elderly. BMC Infect Dis. 2019 Jul 23;19(1):656. doi: 10.1186/s12879-019-4214-x. PMID 31337344
- [Derived] Akmatov MK, Jentsch L, Riese P, May M, Ahmed MW, Werner D, Rosel A, Prokein J, Bernemann I, Klopp N, Prochnow B, Illig T, Schindler C, Guzman CA, Pessler F. Motivations for (non)participation in population-based health studies among the elderly - comparison of participants and nonparticipants of a prospective study on influenza vaccination. BMC Med Res Methodol. 2017 Feb 2;17(1):18. doi: 10.1186/s12874-017-0302-z. PMID 28148221